CLINICAL TRIAL: NCT01856920
Title: A Phase 2 Study of GI-6207 in Patients With Recurrent Medullary Thyroid Cancer
Brief Title: QUILT-3.006 for Recurrent Medullary Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NantCell, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-3.006; 13-C-0095
Record Dates: First submitted 2013-05-08; First posted 2013-05-20 (Estimated); Results first posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Medullary Thyroid Cancer (MTC)
Keywords: Calcitonin; T-cells; Immune Response; HLA Patients; Vaccine
MeSH Terms: conditions — Carcinoma, Medullary | interventions — yeast-CEA vaccine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- A (Experimental): GI-6207 for 1 year
  Interventions: Biological: GI-6207 [Recombinant Saccharomyces cerevisiae-CEA (610D)]
- B (Experimental): 6 months of surveillance followed by GI-6207 for 1 year
  Interventions: Biological: GI-6207 [Recombinant Saccharomyces cerevisiae-CEA (610D)]

INTERVENTIONS:
Biological: GI-6207 [Recombinant Saccharomyces cerevisiae-CEA (610D)] — GI-6207 is a heat-killed, recombinant yeast-based vaccine engineered to express the full length human carcinoembryonic antigen (CEA), with a modified gene coding sequence to code for a single amino acid substitution (asparagine to aspartic acid) at the native protein amino acid position 610, which is designed to enhance immunogenicity. A plasmid vector containing the modified human CEA gene is used to transfect the parental yeast strain (S. cerevisiae W303 - a haploid strain with known mutations from wild-type yeast) to produce the final recombinant vaccine product.

SUMMARY:
Background:

- GI-6207 is an experimental cancer vaccine made with baker's yeast. The yeast has been modified to help the immune system target a protein called CEA. CEA is found on the surface of some kinds of tumor cells, including thyroid cancer cells. Researchers want to see if GI-6207 can encourage the body's immune system to attack and kill tumor cells that contain the CEA protein. They will test to see whether this vaccine is a safe and effective treatment for medullary thyroid cancer that has not responded to earlier treatments.

Objectives:

- To test the safety and effectiveness of the GI-6207 vaccine for advanced medullary thyroid cancer.

Eligibility:

- Individuals at least 18 years of age who have medullary thyroid cancer that has not responded to earlier treatments.

Design:

* Participants will be screened with a physical exam and medical history. They will provide blood and tumor samples and have an imaging study of the neck and chest. They will also have a skin test to make sure that they are not allergic to the yeast in the vaccine.
* Participants will be divided into two groups. One group will start to take GI-6207 immediately for 1 year. The second group will have 6 months of monitoring and tests with no vaccine, and then will take GI-6207 for 1 year.
* GI-6207 will be given every other week for the first seven visits (about 3 months), and then monthly for the remaining year of treatment. It will be given as injections beneath the arm and in the upper thigh. These locations will help the vaccine enter the lymph nodes and reach the immune system more quickly.
* Participants will be monitored with frequent blood and urine tests and imaging studies.
* Participants will have regular follow-up visits after their year of study vaccines.

DETAILED DESCRIPTION:
BACKGROUND:

* CEA is overexpressed in multiple malignancies, including medullary thyroid cancer where CEA is universally expressed on tumor cells.
* There is no standard treatment for patients with asymptomatic or minimally symptomatic, metastatic medullary thyroid cancer. The only effective FDA-approved therapy (vandetanib) comes with significant toxicity, so it is not used until patients have symptomatic or rapidly progressing disease.
* Preclinical studies have shown that GI-6207 can induce a strong immune response to CEA as well as therapeutic anti-tumor responses.
* A previous Phase I GI-6207 study has demonstrated safety and enhanced immune response in some patients.
* Preliminary data suggests that tumor growth rates can be calculated in medullary thyroid cancer patients within 3 months
* Retrospective data from prostate cancer studies suggest that vaccines can alter tumor growth rates within 3-4 months

OBJECTIVES:

Primary:

-To determine the effect of GI-6207 on calcitonin growth rate kinetics after 6 months of therapy in patients with medullary thyroid cancer

ELIGIBILITY:

* Patients will have evidence of metastatic medullary thyroid cancer including disease that is evaluable on bone or CT scan.
* Patients with minimal or no disease related-symptoms (minimal symptoms will include those that do not affect activities of daily living or pain that does not require regularly schedule narcotics.)
* ECOG 0-1
* No previous chemotherapy
* No previous vandetanib
* Should have no autoimmune diseases; no evidence of being immunocompromised; no serious inter-current medical illness; no cardiac disease; no prior splenectomy. (History of previous thyroid autoimmune disease will be allowed as these patients will have had total thyroidectomy.)
* No brain metastasis, history of seizures, encephalitis, or multiple sclerosis
* No pericardial-based masses greater than 1 cm or thoracic lesions larger than 2 cm

Design:

* Randomized, phase 2 study to determine the effect of GI-6207 on calcitonin growth rate after 6 months of GI-6207
* Patients will be randomized to either initial GI-6207 therapy or 6 months of surveillance followed by GI-6207 therapy.
* GI-6207 will be administered subcutaneously at 4 sites at dose of 10 yeast units per site, biweekly for 7 visits (day 1, 15, 29, 43, 57, 71, 85), then monthly up to 1 year of treatment. (For patients randomized to surveillance and then GI-6207, they will get a full year of GI-6207 after a 6 month surveillance period.)
* Once patients have completed one year of therapy with GI-6207, patients without radiographic progression will have the option to receive vaccine every 3 months for an additional 12 months. Patients who remain on vaccine will continue to be scanned every 3 months.
* Immune monitoring via apheresis will be done prior to enrollment and at 6 months for all appropriate and consenting patients. Patients who are evaluable for immunologic response by the ELISPOT Assay (HLA 02, 03 and 24) will have apheresis at start of GI-6207 therapy and then every 3 months while on GI-6207 treatment when feasible.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants must meet the following criteria for participation:

* Diagnosis: Patients must have histologically confirmed medullary thyroid cancer by the Laboratory of Pathology or a pathology report and history consistent with medullary thyroid cancer. It is not uncommon for a secondary, minor pathologic focus of another form of thyroid cancer to be coincidentally found in 15-20% of patients with medullary thyroid cancer. In such cases, eligibility is based on the discretion of the investigator.
* Patients must have evidence of metastatic medullary thyroid cancer including disease that is evaluable on bone, CT scan or MRI. (Patients who are surgical candidates and potentially rendered disease free with surgical resection are not eligible.)
* Patients must have elevated calcitonin levels, greater than 8 pg/mL in females and 16 pg/mL in males
* Patients with minimal or no disease related-symptoms (Minimal symptoms will include those that do not affect activities of daily living or pain that does not require regularly scheduled narcotics.)
* No brain metastasis, history of seizures, encephalitis, or multiple sclerosis.
* Age greater than or equal to 18 years
* ECOG performance status of 0-1 at study entry (Karnofsky greater than or equal to 70)
* No systemic steroid use within 2 weeks prior to initiation of experimental therapy. Limited doses of systemic steroids to prevent IV contrast, allergic reaction or anaphylaxis (in patients who have known contrast allergies) are allowed.
* Hematological eligibility parameters

  * Granulocyte count greater than or equal to 1,500/mm^3
  * Platelet count greater than or equal to 100,000/mm^3
  * Hemoglobin greater than or equal to 9 g/dL
* Biochemical eligibility parameters (within 16 days of starting therapy)

  * Baseline renal function:

    --- Serum creatinine less than or equal to 1.5 x upper limit of normal OR creatinine clearance on a 24-h urine collection of greater than or equal to 60 mL/min.
  * Hepatic function:

    * Bilirubin less than or equal to 1.5 mg/dl, in patients with Gilbert's syndrome, a total bilirubin less than or equal to 3.0 mg/dL
    * AST and ALT< 2.5 times upper limit of normal
* No other active malignancies within the past 3 years (with the exception of nonmelanoma skin cancers, prostate cancer patients with stable biochemical recurrence/not on systemic therapy or carcinoma in situ of the bladder).
* Willing to travel to the NIH for follow-up visits
* Able to understand and sign informed consent.
* Must agree to use effective birth control (such as a condom) or abstinence during and for a period of 6 months after the last vaccination therapy.

EXCLUSION CRITERIA:

Patients with any of the following will not be eligible for participation in this study:

* Patients should have no evidence of immune dysfunction as listed below.

  * 1 Human immunodeficiency virus (HIV) positivity due to the potential for decreased immune response to the vaccine.
  * Active autoimmune diseases requiring treatment or a recent history of autoimmune disease requiring therapy, including, but not limited to, inflammatory bowel disease, Crohn's disease, ulcerative colitis, or active diverticulitis. This requirement is due to the potential risks of exacerbating autoimmunity. However, patients with vitiligo may be enrolled. (Patients with history of autoimmune thyroid conditions will be allowed as these patients will be on replacement medications.)
  * Concurrent use of systemic steroids, except for physiologic doses of systemic steroid replacement or local (topical, nasal, eye drops or inhaled) steroid use. Limited doses of systemic steroids (e.g., in patients with exacerbations of reactive airway disease or to prevent IV contrast allergic reaction or anaphylaxis in patients who have known contrast allergies) are allowed.
* Pregnant or breast-feeding women, due to the unknown effects of GI-6207 on the fetus or infant.
* Serious inter-current medical illness which would interfere with the ability of the patient to carry out the treatment program.
* Untreated brain metastases (or local treatment of brain metastases within the last 6 months) due to the poor prognosis of these patients and difficulty ascertaining the cause of neurologic toxicities.
* Patients with pericardial masses >1 cm or thoracic lesions larger than 2 cm will be excluded.
* Concurrent chemotherapy.
* Chronic hepatitis infection, including B and C, because potential immune impairment caused by these disorders may diminish the effectiveness of this immunologic therapy.
* Participation in another interventional clinical trial at the time of enrollment.
* Any significant disease that, in the opinion of the investigator, may impair the patient's tolerance of study treatment.
* Significant dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
* Patients with second malignancy within 3 years of enrollment; patients treated surgically with a curative intent, such as non-melanoma skin cancers, localized kidney cancer or carcinoma in situ of the bladder, are not excluded. Patients with MEN2 and a history of pheochromocytoma will also not be excluded. In addition patients with prostate cancer who do not require systemic therapy will not be excluded. (A secondary, minor pathologic focus of another form of thyroid cancer may be coincidentally found in 15-20% of patients with medullary thyroid cancer. In such cases, eligibility is based on the discretion of the investigator.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-03-26 (Actual); Primary Completion 2018-05-08 (Actual); Study Completion 2018-05-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- NIH Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Peshwa MV, Shi JD, Ruegg C, Laus R, van Schooten WC. Induction of prostate tumor-specific CD8+ cytotoxic T-lymphocytes in vitro using antigen-presenting cells pulsed with prostatic acid phosphatase peptide. Prostate. 1998 Jul 1;36(2):129-38. doi: 10.1002/(sici)1097-0045(19980701)36:23.0.co;2-d. PMID 9655265
- [Background] Fong L, Small EJ. Anti-cytotoxic T-lymphocyte antigen-4 antibody: the first in an emerging class of immunomodulatory antibodies for cancer treatment. J Clin Oncol. 2008 Nov 10;26(32):5275-83. doi: 10.1200/JCO.2008.17.8954. Epub 2008 Oct 6. PMID 18838703
- [Background] O'Day SJ, Hamid O, Urba WJ. Targeting cytotoxic T-lymphocyte antigen-4 (CTLA-4): a novel strategy for the treatment of melanoma and other malignancies. Cancer. 2007 Dec 15;110(12):2614-27. doi: 10.1002/cncr.23086. PMID 18000991
- [Derived] Del Rivero J, Donahue RN, Marte JL, Gramza A, Bilusic M, Cordes L, Karzai F, Schlom J, Gulley JL, Madan RA. A phase 2 study of GI-6207 in patients with recurrent medullary thyroid cancer. Oncologist. 2025 Dec 30:oyaf429. doi: 10.1093/oncolo/oyaf429. Online ahead of print. PMID 41467761
- [Derived] Del Rivero J, Donahue RN, Marte JL, Gramza AW, Bilusic M, Rauckhorst M, Cordes L, Merino MJ, Dahut WL, Schlom J, Gulley JL, Madan RA. A Case Report of Sequential Use of a Yeast-CEA Therapeutic Cancer Vaccine and Anti-PD-L1 Inhibitor in Metastatic Medullary Thyroid Cancer. Front Endocrinol (Lausanne). 2020 Aug 7;11:490. doi: 10.3389/fendo.2020.00490. eCollection 2020. PMID 32849281
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-C-0095.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Surveillance Subjects: GI-6207 for 1 year
  GI-6207 [Recombinant Saccharomyces cerevisiae-CEA (610D)]: GI-6207 is a heat-killed, recombinant yeast-based vaccine engineered to express the full length human carcinoembryonic antigen (CEA), with a modified gene coding sequence to code for a single amino acid substitution (asparagine to aspartic acid) at the native protein amino acid position 610, which is designed to enhance immunogenicity. A plasmid vector containing the modified human CEA gene is used to transfect the parental yeast strain (S. cerevisiae W303 - a haploid strain with known mutations from wild-type yeast) to produce the final recombinant vaccine product.
- Vaccine Subjects: 6 months of surveillance followed by GI-6207 for 1 year
  GI-6207 [Recombinant Saccharomyces cerevisiae-CEA (610D)]: GI-6207 is a heat-killed, recombinant yeast-based vaccine engineered to express the full length human carcinoembryonic antigen (CEA), with a modified gene coding sequence to code for a single amino acid substitution (asparagine to aspartic acid) at the native protein amino acid position 610, which is designed to enhance immunogenicity. A plasmid vector containing the modified human CEA gene is used to transfect the parental yeast strain (S. cerevisiae W303 - a haploid strain with known mutations from wild-type yeast) to produce the final recombinant vaccine product.
Period: Overall Study
Arm/Group | Surveillance Subjects | Vaccine Subjects
Started | 17 | 18
Completed | 7 | 9
Not Completed | 10 | 9
Not completed — Disease Progression On Study | 3 | 4
Not completed — Disease Progression before Treatment | 1 | 0
Not completed — Ineligible | 0 | 1
Not completed — Patient Declined to Participate (before treatment started.) | 1 | 0
Not completed — Refused further Treatment | 5 | 1
Not completed — Other Reasons | 0 | 1
Not completed — Completed treatment phase but refused the Protocol-Specified | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Surveillance Subjects | Vaccine Subjects | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (14.50) | 51.9 (14.20) | 51.7 (14.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 13 | 13 | 26
  Unknown or Not Reported | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 13 | 13 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6
Patients with recurrent metastatic medullary thyroid cancer [Count of Participants; unit: Participants] | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Calcitonin Growth Rate
Description: NCI developed an equation based on the assumption that the change of a tumor's quantity during therapy results from 2 independent component processes: an exponential (first-order kinetics) decrease/regression and an exponential regrowth of the tumor. The equation is f(t) = exp(-d*t)+exp(g*t) (A) where exp is the base of the natural logarithm, and f(t) is the MTC calcitonin measurement at time t in days, divided by the tumor measurement at day 0, the time at which treatment is commenced. Rate decay constant d (days^(-1) )represents the exponential decrease of the tumor marker signal during therapy. Rate growth constant g (days-^(1) )represents the exponential growth of the tumor during treatment. For each patient an attempt to fit Equation (A) to each data set for which more than one data point is available. Linear regressions to evaluate the relationship between the growth rate constant,g, or other parameters will be implemented using the polynomial linear routine of Sigmaplot 9.0.
Time Frame: after 6 months of therapy
Population: Intent-to-treat: all subjects enrolled in the study regardless of having received treatment
Measure: Number; unit: days^-1
Arm/Group | Surveillance Subjects | Vaccine Subjects
Number analyzed (Participants) | 17 | 18
days^-1 | -2.53 | -2.49
Statistical Analysis 1: Comparison: Surveillance Subjects vs Vaccine Subjects; Test type: Equivalence — Alpha= 0.05; p = 0.3760, Rank-Sum

ADVERSE EVENTS:
Time Frame: All adverse events, including clinically significant abnormal findings on laboratory evaluations, regardless of severity, were to be followed until return to baseline or stabilization of event (up to 2 years). Serious adverse events that occurred more than 30 days after the last administration of investigational agent/intervention and have an attribution of at least possibly related to the agent/intervention were to be recorded (Up to 2 years)
Description: The safety population was used for all adverse event summaries (serious adverse events and non-serious adverse events). Only 13/17 surveillance subjects and 17/18 vaccine subjects received at least one dose of study drug and were included in the safety population.
Arm/Group | Surveillance Subjects | Vaccine Subjects
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/13 | 3/17
Other Adverse Events (participants affected / at risk) | 13/13 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Surveillance Subjects (N=13) | Vaccine Subjects (N=17)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck edema (General disorders) | 0 | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Surveillance Subjects (N=13) | Vaccine Subjects (N=17)
Injection site reaction (General disorders) | 12 | 14
Fatigue (General disorders) | 9 | 8
Flu like symptoms (General disorders) | 4 | 6
Pain (General disorders) | 4 | 6
Fever (General disorders) | 1 | 3
Neck edema (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 7 | 10
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 6
Hypernatremia (Metabolism and nutrition disorders) | 1 | 5
Hyperuricemia (Metabolism and nutrition disorders) | 2 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 4
Hypokalemia (Metabolism and nutrition disorders) | 1 | 4
Hyponatremia (Metabolism and nutrition disorders) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 5 | 9
Nausea (Gastrointestinal disorders) | 4 | 8
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Vomiting (Gastrointestinal disorders) | 2 | 3
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 2
Bloating (Gastrointestinal disorders) | 2 | 0
Constipation (General disorders) | 1 | 1
Stomach pain (Gastrointestinal disorders) | 1 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Oral hemorrhage (Gastrointestinal disorders) | 0 | 1
Lymphocyte count decreased (Investigations) | 4 | 6
Aspartate aminotransferase increased (Investigations) | 3 | 4
Alanine aminotransferase increased (Investigations) | 1 | 5
Creatinine increased (Investigations) | 3 | 2
White blood cell decreased (Investigations) | 1 | 4
CPK increased (Investigations) | 0 | 4
Platelet count decreased (Investigations) | 2 | 2
Alkaline phosphatase increased (Investigations) | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 2
Lipase increased (Investigations) | 0 | 1
Serum amylase increased (Investigations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 4 | 8
Urinary tract infection (Infections and infestations) | 2 | 2
Sinusitis (Infections and infestations) | 1 | 2
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 0 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 2
Amnesia (Nervous system disorders) | 0 | 2
Paresthesia (Nervous system disorders) | 1 | 1
Facial muscle weakness (Nervous system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 2 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 2
Fracture (Injury, poisoning and procedural complications) | 2 | 2
Bruising (Injury, poisoning and procedural complications) | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 3
Anxiety (Psychiatric disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Flushing (Vascular disorders) | 0 | 1
Vascular disorders - Other, specify (Vascular disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 2
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Eye disorders - Other, specify (Eye disorders) | 1 | 0
Flashing lights (Eye disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT01856920/Prot_SAP_000.pdf